CLINICAL TRIAL: NCT07100327
Title: Randomized Controlled Trial (RCT) of Banded Versus Non-Banded Sleeve Gastrectomy in Class IV Obese Patients: 3-Year Follow-up
Brief Title: Banded Versus Non-Banded Sleeve in Class IV Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Professor of General surgery, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT Banded vs Non in Class IV
Record Dates: First submitted 2025-07-17; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Morbid Obesity Requiring Bariatric Surgery
Keywords: Class IV Obese Patients; Banded versus Non-Banded Sleeve Gastrectomy
MeSH Terms: interventions — Chromosome Banding; Chloride-Bicarbonate Antiporters

STUDY DESIGN:
Intervention Model Description: * Banded Group: Laparoscopic sleeve gastrectomy with the placement of a 1.5 x 5.5 cm polypropylene band around the proximal gastric pouch to enhance restriction.
  * Non-Banded Group: Standard laparoscopic sleeve gastrectomy where approximately 75-80% of the stomach is resected to form a tubular structure.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Banded Group (Active Comparator): Placement of a 1.5 x 5.5 cm polypropylene band
  Interventions: Procedure: Band
- Non-Banded Group (Placebo Comparator): Standard laparoscopic sleeve gastrectomy
  Interventions: Procedure: Non-Band

INTERVENTIONS:
Procedure: Band — Laparoscopic sleeve gastrectomy with the placement of a 1.5 x 5.5 cm polypropylene band around the proximal gastric pouch to enhance restriction.
  Arms: Banded Group
Procedure: Non-Band — Standard laparoscopic sleeve gastrectomy where approximately 75-80% of the stomach is resected to form a tubular structure
  Arms: Non-Banded Group

SUMMARY:
Obesity remains a major global health challenge, with Class IV super obesity (BMI ≥ 50 kg/m²) being the most severe form. This condition is associated with numerous comorbidities including type 2 diabetes, hypertension, obstructive sleep apnea, and hyperlipidemia, which significantly reduce life expectancy and quality of life. Bariatric surgery, particularly sleeve gastrectomy (SG), has been shown to be an effective treatment for morbid obesity. While SG results in significant weight loss and improvement of comorbidities, some patients experience weight regain over time.

Banded sleeve gastrectomy (BSG) has been proposed as a modification of SG to enhance long-term outcomes by providing additional restriction via a polypropylene band around the proximal gastric pouch. Although initial evidence for banded procedures suggests improved outcomes, particularly in the context of weight loss and reduced weight regain, specific evidence for Class IV obesity remains limited.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of adding a band to sleeve gastrectomy in patients with Class IV obesity by comparing weight loss, comorbidity resolution, complications, and quality of life outcomes over a 3-year period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years
* BMI ≥ 50 kg/m² (Class IV obesity)
* No prior gastrointestinal surgeries
* No significant psychiatric or medical contraindications to surgery
* Ability to provide informed consent

Exclusion Criteria:

* BMI < 50 kg/m²
* Refusal to undergo band placement
* Active reflux disease or PPI use
* Prior bariatric surgery
* Pregnancy plans during the study period
* Active cancer or life-limiting illness
* Substance abuse or non-compliance with postoperative care
* Gastroesophageal reflux disease.
* Hiatal hernia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 219 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Total Weight Loss (TWL) | Measured at 6, 12, 24 and 36 months postoperatively
  Total Weight Loss between the 2 groups (in kilograms)

SECONDARY OUTCOMES:
Resolution of associated medical problems | 6, 12, 24, and 36 months.
  Improvement or resolution of conditions like type 2 diabetes. Your doctor or a healthcare professional will perform a simple blood test, which may involve a finger prick or drawing blood from your arm.
  If a finger prick is used, you may get immediate results. If blood is sent to a lab, results are typically available within a day.
  The HbA1c (Hemoglobin A1c) test is a blood test used to measure your average blood sugar (glucose) levels over the past two to three months, providing a long-term indicator of blood glucose control and helping to diagnose and monitor diabetes and prediabetes.
  An HbA1c level below 5.7% is considered healthy. A result between 5.7% and 6.4% indicates prediabetes. A result of 6.5% or higher on two separate tests is used to diagnose diabetes. For individuals with diabetes, the HbA1c test helps monitor the effectiveness of diabetes management.
Resolution of associated medical problems | 6, 12, 24, and 36 months.
  Improvement or resolution of conditions like hypertension. Blood pressure is measured in millimeters of mercury (mmHg) and is expressed as two numbers: systolic pressure (when the heart beats) over diastolic pressure (when the heart rests). A normal blood pressure reading is generally considered to be below 120/80 mmHg.
  Normal Blood Pressure: Generally, a reading of 120/80 mmHg or lower is considered normal.
  High Blood Pressure (Hypertension): Readings of 130/80 mmHg or higher are generally considered high.
Resolution of associated medical problems | 6, 12, 24, and 36 months.
  Improvement or resolution of conditions like obstructive sleep apnea. Obstructive Sleep Apnea (OSA) severity is primarily measured using the Apnea-Hypopnea Index (AHI), which quantifies the number of breathing interruptions (apneas) and reduced airflow episodes (hypopneas) per hour of sleep. The AHI, determined through polysomnography (PSG), categorizes OSA as mild (AHI 5-14), moderate (AHI 15-30), or severe (AHI >30).
Resolution of associated medical problems | 6, 12, 24, and 36 months.
  Improvement or resolution of conditions like hyperlipidemia. Hyperlipidemia, or high cholesterol, is measured through a lipid panel, a blood test that assesses various types of cholesterol and triglycerides, with results typically reported in milligrams per deciliter (mg/dL). This test usually requires a period of fasting beforehand, and a healthcare professional will draw a blood sample from a vein.
Complications | post operative, 12, 24, and 36 months
  Postoperative complications classified by the Clavien-Dindo system.
Food Intolerance | 12, 24, and 36 months
  Measured through patient-reported outcomes using the validated food intolerance questionnaire by Suter et al.
Volumetric Analysis | 12, 24, and 36 months
  Evaluation of the gastric pouch volume postoperatively using radiographic imaging or endoscopic techniques
Quality of Life (QOL) | 6, 12, 24, and 36 months
  Assessed using validated questionnaires such as the SF-36
BODY-Q | 12, 24, and 36 months
  Assessed using validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ashour, Ph.D. (Professor), Principal Investigator — The surgical department of Medical Research Institute Hospital, Alexandria University
Locations (1):
- The surgical department of Medical Research Institute Hospital, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The analysis will be performed on a blinded dataset after completing the medical/scientific review. All protocol violations will be identified and resolved, and the dataset will be declared complete. All data will be collected in a data management system (Castor EDC, Amsterdam, The Netherlands; https://www.castoredc.com), handled according to Good Clinical Practice guidelines, Data Protection Directive certificate, and complied with Title 21 CFR Part 11. Furthermore, the data centers where all the research data will be stored are certified according to ISO27001, ISO9001, and Dutch NEN7510.
  Can be asked by the contact person
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: whole study period
Access Criteria: Ask contact person